CLINICAL TRIAL: NCT03022370
Title: Stepping Stones and Creating Futures Intervention Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of KwaZulu (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Department for International Development, United Kingdom (Other Government); Project Empower (Other)
Responsible Party: Principal Investigator, Andrew Gibbs, Principal Investigator, Senior Specialist Scientist, Medical Research Council, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BFC043/15
Record Dates: First submitted 2017-01-05; First posted 2017-01-16 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: IPV; Sexual Violence
Keywords: informal settlements; poverty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepping Stones and Creating Futures (Experimental): Participants receive the Stepping Stones and Creating Futures intervention, comprising of 21 participatory/inter-active sessions, delivered by a trained facilitators. Each session last approximately 3 hours. Sessions are delivered twice a week. Sessions are primarily single sex, with 20 participants per group.
  Interventions: Behavioral: Stepping Stones and Creating Futures
- Wait-list control (No Intervention): Participants receive no intervention until after final data collection occurs, at which point they will be offered Stepping Stones and Creating Futures.

INTERVENTIONS:
Behavioral: Stepping Stones and Creating Futures — Stepping Stones consists of 10 sessions. It seeks to strengthen relationships and to transform views on gender and in the process impact on exposure to, or participation in, gender-based violence and HIV risk. These cover gender and peer influences our actions; sex and love; conception and contraception; STIs and HIV; safer sex and condoms; GBV; motivations for behaviour (including influences of alcohol and poverty); and communication skills.
  Creating Futures is a facilitated group intervention of eleven sessions. It seeks to strengthen livelihoods. The key sessions include: setting medium term livelihood goals, the need for assets and coping with crises; social resources for livelihoods (trust and community participation); getting and keeping jobs; and savings and spending.
  Arms: Stepping Stones and Creating Futures

SUMMARY:
This study evaluates whether the behavioural/structural interventions of Stepping Stones and Creating Futures can reduce the incidence of intimate partner violence in urban informal settlements amongst young people. Half the participants will receive the interventions, while the other half will be in a control wait-list, only receiving the intervention after final data collection.

ELIGIBILITY:
Inclusion Criteria:

* Normally resident in informal settlement cluster
* Not formally employed
* Able to communicate in main study languages (English, isiZulu, iXhosa)

Exclusion Criteria:

* Under 18
* Mental deficit (learning difficulty, mental illness or substance abuse)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1351 (Actual)
Dates: Start 2015-10; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gibbs, PhD, Principal Investigator — Gender and Health Research Unit, South African Medical Research Council (SAMRC); Health Economics and HIV/AIDS Research Division (HEARD), University of KwaZulu Natal
Locations (1):
- Gender and Health Research Unit, South African Medical Research Council, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibbs A, Washington L, Willan S, Ntini N, Khumalo T, Mbatha N, Sikweyiya Y, Shai N, Chirwa E, Strauss M, Ferrari G, Jewkes R. The Stepping Stones and Creating Futures intervention to prevent intimate partner violence and HIV-risk behaviours in Durban, South Africa: study protocol for a cluster randomized control trial, and baseline characteristics. BMC Public Health. 2017 Apr 20;17(1):336. doi: 10.1186/s12889-017-4223-x. PMID 28427380
- [Background] Gibbs A, Dunkle K, Washington L, Willan S, Shai N, Jewkes R. Childhood traumas as a risk factor for HIV-risk behaviours amongst young women and men living in urban informal settlements in South Africa: A cross-sectional study. PLoS One. 2018 Apr 6;13(4):e0195369. doi: 10.1371/journal.pone.0195369. eCollection 2018. PMID 29624612
- [Background] Gibbs A, Dunkle K, Jewkes R. Emotional and economic intimate partner violence as key drivers of depression and suicidal ideation: A cross-sectional study among young women in informal settlements in South Africa. PLoS One. 2018 Apr 16;13(4):e0194885. doi: 10.1371/journal.pone.0194885. eCollection 2018. PMID 29659595
- [Background] Gibbs A, Washington L, Abdelatif N, Chirwa E, Willan S, Shai N, Sikweyiya Y, Mkhwanazi S, Ntini N, Jewkes R. Stepping Stones and Creating Futures Intervention to Prevent Intimate Partner Violence Among Young People: Cluster Randomized Controlled Trial. J Adolesc Health. 2020 Mar;66(3):323-335. doi: 10.1016/j.jadohealth.2019.10.004. Epub 2019 Nov 26. PMID 31784410
- [Derived] Gibbs A, Mkhwanazi S, Khaula S, Washington L, Sikweyiya Y. A Prospective Analysis of Associations Between Changes in Mental Health and Men's Perpetration of Intimate Partner Violence: Post-Hoc Analysis of Young Men Involved in the Stepping Stones and Creating Futures Trial. J Interpers Violence. 2026 Jan 21:8862605251408126. doi: 10.1177/08862605251408126. Online ahead of print. PMID 41562393
- [Derived] Oyekunle V, Gibbs A, Tomita A. Assessing the role of depression in reducing intimate partner violence perpetration among young men living in urban informal settlements using a mediation analysis of the Stepping Stones and Creating Futures intervention. Glob Health Action. 2023 Dec 31;16(1):2188686. doi: 10.1080/16549716.2023.2188686. PMID 36927500
- [Derived] Mannell J, Minckas N, Burgess R, Chirwa ED, Jewkes R, Gibbs A. Does experiencing a traumatic life event increase the risk of intimate partner violence for young women? A cross-sectional analysis and structural equation model of data from the Stepping Stones and Creating Futures intervention in South Africa. BMJ Open. 2022 Apr 29;12(4):e051969. doi: 10.1136/bmjopen-2021-051969. PMID 35487735
- [Derived] Gibbs A, Dunkle K, Mhlongo S, Chirwa E, Hatcher A, Christofides NJ, Jewkes R. Which men change in intimate partner violence prevention interventions? A trajectory analysis in Rwanda and South Africa. BMJ Glob Health. 2020 May;5(5):e002199. doi: 10.1136/bmjgh-2019-002199. PMID 32424011
- [Derived] Gibbs A, Jewkes R, Willan S, Washington L. Associations between poverty, mental health and substance use, gender power, and intimate partner violence amongst young (18-30) women and men in urban informal settlements in South Africa: A cross-sectional study and structural equation model. PLoS One. 2018 Oct 3;13(10):e0204956. doi: 10.1371/journal.pone.0204956. eCollection 2018. PMID 30281677

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stepping Stones and Creating Futures | Wait-list Control
Started | 677 | 674
Completed | 497 | 553
Not Completed | 180 | 121
Not completed — Death | 6 | 12
Not completed — Lost to Follow-up | 174 | 109

BASELINE CHARACTERISTICS:
Groups:
- Women - Intervention: Women who received the Stepping Stones and Creating Futures intervention
- Men - Intervention: Men who received the intervention
- Women - Control: Women in the wait list control
- Men - Control: Men in the wait list control
- Total: Total of all reporting groups
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control | Total
Number analyzed (Participants) | 339 | 338 | 338 | 336 | 1351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 339 | 338 | 338 | 336 | 1351
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 339 | 0 | 338 | 0 | 677
  Male | 0 | 338 | 0 | 336 | 674
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Africa | 339 | 338 | 338 | 336 | 1351

OUTCOME MEASURES:

1. Primary Outcome: Any Past Year Physical Intimate Partner Violence Perpetration (Men) and Experience (Women)
Description: Physical intimate partner violence is assessed using five items based on the WHO VAW scale. A positive response to any item leads to a person being classified as perpetrating (men) and experiencing (women) in the past year. With 0=none, 1=yes.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Participants | 134 | 86 | 155 | 118
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.686, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.62 to 1.37]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.51 to 0.97]

2. Primary Outcome: Any Past Year Sexual Intimate Partner Violence Perpetration (Men) and Experience (Women)
Description: Sexual intimate partner violence is assessed using three items based on the WHO VAW scale. A positive response to any item leads to a person being classified as perpetrating (men) and experiencing (women) in the past year. With 0=none, 1=yes.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Participants | 86 | 52 | 101 | 73
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.555, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.64 to 1.28]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.072, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.54 to 1.03]

3. Primary Outcome: Past Year Severe Sexual and/or Physical Intimate Partner Violence Perpetration (Men) and Experience (Women)
Description: Severe sexual and/or physical intimate partner violence perpetration (men) and experience (women) is assessed using 8 items. Past year severe sexual and/or physical IPV is assessed as positive if a person responds to two (or more) items as once, or one item as few (or more), essentially creating a more than once categorization.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Participants | 151 | 99 | 171 | 135
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.672, Regression, Logistic; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.66 to 1.31]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.019, Regression, Logistic; Odds Ratio (OR) = 0.70, 95% CI 2-sided [0.52 to 0.94]

4. Primary Outcome: Controlling Behaviours
Description: Controlling behaviours are assessed using a modified Sexual Relationship Power (SRP) scale. Men's control of female sexual partner's and women's experience of controlling behaviours from a male partner. A mean score is calculated with higher scores indicating more controlling (bad). Range: 0-24
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 9.75 [9.17 to 10.32] | 9.96 [9.36 to 10.56] | 9.70 [9.12 to 10.22] | 9.96 [9.44 to 10.47]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.984, Regression, Linear; Slope = -0.01, 95% CI 2-sided [-0.88 to 0.86]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.839, Regression, Linear; Slope = 0.06, 95% CI 2-sided [-0.51 to 0.63]

5. Primary Outcome: Earnings in Past Month
Description: A single item question asks "Considering all the money you earned from jobs or selling things (excluding grants), how much did you earn last month?" Responses are in Rands and a continuous scale, with no upper limit.
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: Rands
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Rands | 565 [443 to 688] | 988 [798 to 1177] | 385 [268 to 503] | 817 [594 to 1038]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p < 0.0001, Tobit; Log + 1 performed on data; Slope = 0.97, 95% CI 2-sided [0.43 to 1.51]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.521, Tobit; Log plus 1 to transform data; Slope = 0.21, 95% CI 2-sided [-0.42 to 0.83]

6. Secondary Outcome: Gender Attitudes
Description: Modified gender equitable men's scale (GEMS) assess participant's gender attitudes. A mean score is calculated with higher scores indicative of more gender inequitable attitudes (range: 0-60)
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 21.98 [20.78 to 23.18] | 24.99 [23.58 to 26.39] | 21.65 [20.74 to 22.72] | 25.15 [23.93 to 26.38]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.718, Regression, Linear; Slope = 0.25, 95% CI 2-sided [-1.09 to 1.58]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.712, Regression, Linear; Slope = -0.30, 95% CI 2-sided [-1.87 to 1.28]

7. Secondary Outcome: Depressive Symptomology
Description: Past week depressive symptomology is assessed by the Centre for Epidemiological Studies Depression (CESD) scale, with the full twenty items (range 0-60). A mean score is calculated, with higher scores indicating more depression.
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 21.95 [20.70 to 23.20] | 19.26 [18.06 to 20.47] | 23.11 [21.86 to 24.36] | 20.35 [19.26 to 20.47]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.067, Regression, Linear; Slope = -1.52, 95% CI 2-sided [-3.14 to 0.11]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.398, Regression, Linear; Slope = -0.75, 95% CI 2-sided [-2.48 to 0.99]

8. Secondary Outcome: Number of Participants Reporting Suicidal Ideation
Description: Past four week suicidal ideation was assessed using a single item question. Responses are either 0=no, or 1=yes.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Participants | 83 | 49 | 72 | 65
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.228, Regression, Logistic; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.85 to 1.97]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.558, Regression, Logistic; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.53 to 1.41]

9. Secondary Outcome: Life Circumstances
Description: Four items modified from the Satisfaction with Life Scale (SWLS) by Denier et al. (1985), with items on a five point Likert Scale (range 0-20) higher scores indicative of greater life satisfaction.
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 10.28 [9.82 to 10.75] | 10.59 [10.13 to 11.06] | 9.88 [9.47 to 10.29] | 10.03 [9.62 to 10.43]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.679, Regression, Linear; Slope = 0.14, 95% CI 2-sided [-0.52 to 0.80]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.08, Regression, Linear; Slope = 0.55, 95% CI 2-sided [-0.07 to 1.16]

10. Secondary Outcome: Problem Alcohol Use
Description: Problem drinking in the past year is assessed using the AUDIT (alcohol use disorders identification test) scale. With a range of 0-40, and recoded with scores of 8 or more classifing a participant as having potentially problematic alcohol use.
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 4.27 [3.49 to 5.06] | 6.81 [5.86 to 7.75] | 4.62 [3.80 to 5.45] | 7.97 [6.94 to 8.99]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.810, Regression, Linear; Slope = -0.13, 95% CI 2-sided [-1.21 to 0.95]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.041, Regression, Linear; Slope = -1.03, 95% CI 2-sided [-2.01 to -0.04]

11. Secondary Outcome: Number of People Quarreling With Partner About Alcohol Use
Description: A single item binary response question asks whether participants have argued about alcohol with their sexual partner in the past year (0=no; 1=yes). Only asked to those who reported alcohol use in the past year.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 129 | 160 | 138 | 184
Participants | 39 | 54 | 47 | 79
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.635, Regression, Logistic; Odds Ratio (OR) = 1.14, 95% CI 2-sided [0.67 to 1.92]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.256, Regression, Logistic; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.41 to 1.27]

12. Secondary Outcome: Last Sexual Partner of Participant is the Main Partner
Description: A single item assess who the participant last had sex with, with possible responses being: "main partner", "casual partner", "once-off sex partner" or "ex-partner". As per the protocol, we recategorised this into either "1=main partner" or "0=other". Positive change is towards main partner. And the reported number (proportion) is those reporting Main partner.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 236 | 220 | 243 | 258
Participants | 185 | 138 | 182 | 159
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.526, Regression, Logistic; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.73 to 1.84]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.931, Regression, Logistic; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.67 to 1.56]

13. Secondary Outcome: Transactional Sex Past Year
Description: Five item scale asks about transactional sex with casual or once-off sexual partners in the past year based on the scale developed and tested by Dunkle et al (2004). Each item has a no/yes response. A response of yes to any is classified as having engaged in transactional sex.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 236 | 220 | 243 | 258
Participants | 111 | 138 | 118 | 146
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.691, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.63 to 1.36]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.692, Regression, Logistic; Odds Ratio (OR) = 0.92, 95% CI 2-sided [0.60 to 1.40]

14. Secondary Outcome: Shame About Lack of Work
Description: Four items assess participants' feelings of shame about not enough work, based on a scale developed for use in the IMAGES study, with . Mean score calculated, with higher scores indicative of more shame (range: 4-16)
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 10.3 [9.9 to 10.6] | 10.7 [10.4 to 11.1] | 10.7 [10.4 to 10.9] | 10.9 [10.6 to 11.2]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.137, Regression, Linear; Slope = -0.31, 95% CI 2-sided [-0.72 to 0.24]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.721, Regression, Linear; Slope = -0.09, 95% CI 2-sided [-0.58 to 0.40]

15. Secondary Outcome: Stress About Lack of Work
Description: Four items assess participants' feelings of stress about not enough work, based on a scale developed for the IMAGES study. Mean score calculated, with higher scores indicating more stress (range: 4-20)
Time Frame: 24 months post baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
score on a scale | 12.0 [11.6 to 12.3] | 11.8 [11.5 to 12.2] | 12.1 [11.8 to 12.5] | 12.0 [11.7 to 12.3]
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.332, Regression, Linear; Slope = -0.23, 95% CI 2-sided [-0.70 to 0.24]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.468, Regression, Linear; Slope = -0.19, 95% CI 2-sided [-0.71 to 0.32]

16. Secondary Outcome: Individual's Ability to Mobilise Money in an Emergency
Description: A single item asks participants how hard it would be to mobilise R200 (~US$15) in an emergency. Those responding it would be "very difficult, or somewhat difficult" are classified as finding it hard (=1). Those responding "fairly easy or easy" are classified as not finding it hard (=0). Reported number (proportion) is of those finding it hard to mobilise money in an emergency. A positive change is towards a lower proportion.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Participants | 27 | 37 | 30 | 31
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.174, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.89 to 1.90]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.129, Regression, Logistic; Odds Ratio (OR) = 1.49, 95% CI 2-sided [0.89 to 2.50]

17. Secondary Outcome: Stolen Because of Hunger in Past Month
Description: Single item question asks about stealing because of lack of food or money in the past month with responses "never", "once", "every week" or "every day". Responses are recoded, as per protocol, into "0=never" and "1=once or more". The number/proportion of those stealing in the past month is reported. A lower proportion is a positive change.
Time Frame: 24 months post baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
Number analyzed (Participants) | 260 | 237 | 285 | 268
Participants | 88 | 91 | 84 | 105
Statistical Analysis 1: Comparison: Women - Intervention vs Women - Control; Test type: Superiority; p = 0.174, Regression, Logistic; Odds Ratio (OR) = 1.30, 95% CI 2-sided [0.89 to 1.90]
Statistical Analysis 2: Comparison: Men - Intervention vs Men - Control; Test type: Superiority; p = 0.836, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.64 to 1.43]

ADVERSE EVENTS:
Time Frame: 24 months of follow up
Arm/Group | Women - Intervention | Men - Intervention | Women - Control | Men - Control
All-Cause Mortality (participants affected / at risk) | 5/339 | 3/338 | 3/338 | 7/336
Serious Adverse Events (participants affected / at risk) | 3/339 | 2/338 | 0/338 | 0/336
Other Adverse Events (participants affected / at risk) | 0/339 | 0/338 | 0/338 | 0/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women - Intervention (N=339) | Men - Intervention (N=338) | Women - Control (N=338) | Men - Control (N=336)
Violence experience (Social circumstances) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Participants experienced violence other men
Hospitalisation (Social circumstances) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — We did not collect detailed information on causes of hospitalisation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT03022370/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT03022370/SAP_001.pdf
  • Informed Consent Form (2015-11-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT03022370/ICF_002.pdf